CLINICAL TRIAL: NCT04393662
Title: TenTed-Postoperative Biceps Strength and Electromyographic Activity After Proximal Biceps Tenotomy Versus Tenodesis in Patients With Arthroscopic Rotator Cuff Tear Repair
Brief Title: Postoperative Biceps Strength and Electromyographic Activity After Proximal Biceps Tenotomy Versus Tenodesis in Patients With Arthroscopic Rotator Cuff Tear Repair
Acronym: TenTed
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02004; ch20Taha
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Biceps Tendon Lesion
Keywords: partial rotator cuff tear; complete rotator cuff tear; proximal biceps tenotomy; proximal biceps tenodesis; arthroscopic rotator cuff tear repair; biceps strength in supination and flexion; Supination Strength Index SSI; lesion of the long head of the biceps tendon (LHBT)
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tenodesis group: Tenodesis as surgical treatment option for a lesion of the long head of the biceps tendon (LHBT)
  Interventions: Diagnostic Test: Measurement of Muscle strength using a dynamometer; Diagnostic Test: Range of motion clinical measurement (shoulder and elbow); Diagnostic Test: Electromyography (EMG)
- Tenotomy group: Tenotomy as surgical treatment option for a lesion of the long head of the biceps tendon (LHBT)
  Interventions: Diagnostic Test: Measurement of Muscle strength using a dynamometer; Diagnostic Test: Range of motion clinical measurement (shoulder and elbow); Diagnostic Test: Electromyography (EMG)

INTERVENTIONS:
Diagnostic Test: Measurement of Muscle strength using a dynamometer — Muscle strength will be measured in the elbow bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA). Supination tests will be performed with the forearm in neutral position, 60° pronation and 60° supination. The elbow will be in 90° flexion, and the shoulder in 45° flexion. Constant pressure is applied to lever of device for 3 to 5 seconds. Maximum torque will be recorded automatically. For each position, three repetitions of 3s (to 5s) contractions will be performed with a break of 15 (or 30s) between the repetitions. There will be an additional break of 2 minutes between measurements of the supination strength in the different positions. This parameter will be analysed regarding asymmetry between both limbs.
  Isometric endurance of forearm supination will be measured in neutral forearm. Flexion tests will be carried in the same setting as for supination. Flexion tests will be performed with the elbow in 90, 45 and 0° of flexion.
Diagnostic Test: Range of motion clinical measurement (shoulder and elbow) — The range of motion parameters (degree) of both shoulders and elbows will be documented. The circumference of the arm will be measured on the line between the medial acromion and the cubital fossa at 1/3 from the cubital fossa
Diagnostic Test: Electromyography (EMG) — Electromyographic (EMG) data will be collected using a wireless EMG system (myon AG, Schwarzenberg, Switzerland). Surface electrodes will be placed bilaterally on biceps and triceps following the guidelines of the SENIAM project (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles)

SUMMARY:
The most important functions of the biceps brachii muscle are flexion and supination of the elbow. Patients with a partial or complete rotator cuff tear often suffer a lesion of the long head of the biceps tendon (LHBT). The two most common surgical treatments options are tenotomy or tenodesis. This study is to assess the Supination Strength Index (SSI) (the operated side in relation to the healthy side) after proximal biceps tenotomy versus tenodesis.

DETAILED DESCRIPTION:
The most important functions of the biceps brachii muscle are flexion and supination of the elbow. Patients with a partial or complete rotator cuff tear often suffer a lesion of the long head of the biceps tendon (LHBT). The two most common surgical treatments options are tenotomy or tenodesis. This study is to assess the Supination Strength Index SSI (the operated side in relation to the healthy side) after proximal biceps tenotomy versus tenodesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient after an arthroscopic rotator cuff repair who underwent a biceps tenotomy or tenodesis
* 1-4 years postoperative
* Written informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Previous biceps injury and or operation
* Contralateral biceps injury
* Neurological disorders potentially affecting upper extremity muscle strength.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be asked to participate in clinical and functional analysis after an arthroscopic rotator cuff repair who underwent a biceps tenotomy or tenodesis (1 to 4 years after surgery) at the University Hospital Basel between Jan 2015 and Oct 2018.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Supination Strength Index SSI | at Baseline
  comparison of the Supination Strength Index SSI (the operated side in relation to the healthy side). It is calculated by dividing the strength on the operated side by the strength on the healthy side.

SECONDARY OUTCOMES:
patient's pain visual analog scale Score (VAS) | at Baseline
  patient's pain visual analog scale score (VAS): 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable
American Shoulder and Elbow Surgeons (ASES) Score | at Baseline
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living. Calculation of the ASES score is a complicated process. The final pain score is calculated via an independent formula, while the raw score from the functional questions is multiplied by a coefficient to get the final score for the functional questions. The pain and functional portions are then summed to obtain the final ASES score with higher scores indicating better outcomes
Constant Score | at Baseline
  This scoring system consists of four variables that are used to assess the function of the shoulder. The right and left shoulders are assessed separately.
  The subjective variables are pain and activities of daily living (ADL) (sleep, work, recreation / sport) which give a total of 35 points. The objective variables are range of motion and strength which give a total of 65 points. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
Long head of Biceps Score (LHB-Score) | at Baseline
  The LHB score (maximum 100 points) described by Scheibel et al. evaluates the qualities ''biceps pain and muscle cramps'' (maximum 50 points), ''cosmesis" (maximum 30 points) and ''flexion strength at the elbow'' (maximum 20 points)
muscle activation determined from electromyographic (EMG) data | at Baseline
  The level of muscle activation of the biceps during forearm supination will be expressed as percentage of the peak muscle activation during elbow flexion and compared between the limbs of each patient. The mean frequency of the muscle activation will be calculated using a Fast Fourier Transform in 1s windows. Fatigue will be determined as the change in the mean frequency from the beginning of the endurance task to the end of the endurance task
supination muscle strength | at Baseline
  Isometric endurance of forearm supination will be measured in neutral forearm. Participants will be asked to maximally supinate their forearm for as long as possible. Endurance will be quantified as the elapsed time until the patient stops the measurement due to fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Mueller, PD Dr. med., Principal Investigator — Orthopädie/Traumatologie University Hospital Basel
Locations (1):
- Orthopädie/Traumatologie University Hospital Basel, Basel, Switzerland